CLINICAL TRIAL: NCT07230392
Title: Comparison of Superficial Cervical Plexus Block and Ketamine in the Prevention of Chronic Pain After Thyroidectomy: Results of a Prospective Randomized Study
Brief Title: Superficial Cervical Plexus Block Versus Ketamine in the Prevention of Chronic Pain After Thyroidectomy
Acronym: Thyrobloket
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben Taleb Ibtissem, Assistant Professor in Anesthesiology and Intensive Care, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Thyrobloket
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Thyroidectomy
Keywords: Ketamine; Thyroidectomy; Cervical block
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCS Group (Active Comparator): Patients received a bilateral ultrasound-guided superficial cervical plexus block after induction (Ropivacaine 0.2%,with a volume of 10 mL administered to each side)
  Interventions: Procedure: Superficial cervical plexus block
- KETA group (Active Comparator): Patients received intravenous ketamine (0.25 mg/kg bolus followed by a 2 µg/kg/min infusion).
  Interventions: Drug: Ketamine perfusion

INTERVENTIONS:
Drug: Ketamine perfusion — Intravenous ketamine 0.25 mg/kg bolus followed by a 2 µg/kg/min infusion
  Arms: KETA group
Procedure: Superficial cervical plexus block — Bilateral ultrasound-guided superficial cervical plexus block after induction(Ropivacaine 0.2% Ropivacaine 0.2%, with a volume of 10 mL administered to each side) was performed for patients of this group
  Arms: BCS Group

SUMMARY:
The goal of our work is to to compare the effect of preemptive Ketamine administration versus superficial cervical plexus block on the incidence of postoperative neuropathic pain in patients undergoing thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years
* Scheduled for thyroidectomy under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Able to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Known allergy to ketamine or local anesthetics
* Severe renal impairment with estimated Glomerular Filtration Rate (eGFR) under 30 mL/min
* History of neurological disorders
* History of psychiatric illness
* History of severe cardiac disease (NYHA III-IV) or serious arrhythmias
* Pregnancy or breastfeeding
* Morbid obesity (BMI > 40 kg/m²)
* Cognitive or communication impairment
* Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
The incidence of chronic neuropathic pain at three months | three months after thyroidectomy
  The incidence of chronic neuropathic pain at three months after thyroidectomy, as determined by the DN4 questionnaire.

SECONDARY OUTCOMES:
Twenty-four hour postoperative rescue analgesia requirements | within the first 24 hours after the thyroidectomy.
  The total amount of extra, on-demand pain medication a patient needed in the first 24 hours after their surgery was completed.
Intraoperative sufentanil consumption | During the intraoperative period
  The secondary endpoints included intraoperative sufentanil consumption and reinjection requirements.
Postoperative sleep quality | During the first 24 postoperative hours.
  Sleep quality was assessed 24 hours postoperatively to accurately reflect the effects of analgesia, utilizing the Athens Insomnia Scale (AIS) score.
Incidence of postoperative nausea and vomiting (PONV) within 24 hours post-surgery | 24 hours after surgery.
  Occurrence of at least one episode of nausea or vomiting within the first 24 hours after surgery.
The Observer's Assessment of Alertness/Sedation (OAA/S) within a 2-hour timeframe following thyroidectomy. | 2-hour timeframe following thyroidectomy
  Patients underwent Observer's Assessment of Alertness/Sedation (OAA/S) assessment within a 2-hour timeframe following thyroidectomy, before being cleared for PACU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: ibtissem BEN TALEB, Principal Investigator — University of Tunis El Manar, Anesthesia and critical care department, Taher Maamouri University Hospital,
Locations (1):
- Mohamed Taher Maamouri University Hospital, Nabeul, Nabeul Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided